CLINICAL TRIAL: NCT07083492
Title: Point-of-care Transcutaneous Longitudinal Non-invasive Detection of Iron Deficiency in Obstetrics (PICCOLINO-Trial)
Brief Title: Non-invasive Detection of Iron Deficiency in Obstetrics
Acronym: PICCOLINO
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. P. Kranke, Prof. Dr. P. Kranke, Wuerzburg University Hospital
Other Study IDs: 115/21-sc
Record Dates: First submitted 2022-11-12; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Iron Deficiency Anemia of Pregnancy; Iron-deficiency; Restless Leg Syndrome in Pregnancy; Restless Leg Syndrome Due to Iron Deficiency Anaemia; Postpartum Hemorrhage; Postpartum Depression; Pregnancy Anemia; Iron Deficiency (Without Anemia)
Keywords: Zinc protoporphyrin; Non-invasive detection; Obstetric anesthesia; Patient blood management
MeSH Terms: conditions — Anemia, Iron-Deficiency; Postpartum Hemorrhage; Depression, Postpartum; Iron Deficiencies | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women
  Interventions: Diagnostic Test: non-invasive measurement of zink protoporphyrin

INTERVENTIONS:
Diagnostic Test: non-invasive measurement of zink protoporphyrin — validation of non-invasive measurement of zink protoporphyrin
  Other Names: blood samples; questionnaires

SUMMARY:
Validation of non-invasive measurement of zinc protoporphyrin for detection of iron deficiency in pregnancy.

In addition, the impact of iron deficiency on the incidence of postpartum depression, restless legs syndrome, obstetric complications and quality of life will be examined.

DETAILED DESCRIPTION:
Study Title Point-of-care transcutaneous longitudinal non-invasive detection of iron deficiency in obstetrics (PICCOLINO Trial)

________________________________________ Brief Summary Iron deficiency is a common condition during pregnancy and is associated with maternal fatigue, increased need for blood transfusion during delivery, and adverse neonatal outcomes. However, current screening practices are inconsistent and often rely on imprecise laboratory parameters like hemoglobin and ferritin. The PICCOLINO trial is a prospective, longitudinal observational study investigating the feasibility and diagnostic value of a novel non-invasive fluorescence-based device to measure zinc protoporphyrin (ZnPP) at the lower lip as a screening tool for iron deficiency in pregnant women.

This study compares non-invasive ZnPP measurements with conventional blood-based markers for iron deficiency and anemia at five time points: once in each trimester, at the time of delivery, and approximately 2-3 months postpartum. The study further examines correlations between iron status and maternal well-being, postpartum depression, restless legs syndrome (RLS), and pregnancy complications.

________________________________________ Detailed Description The study enrolls up to 500 pregnant women, aiming to start inclusion as early as the first trimester. In each participant, ZnPP will be measured non-invasively at the lower lip using an optical sensor. Concurrently, venous blood samples will be drawn (where possible during routine care) to assess standard hematological and iron-related parameters (Hb, MCV, MCH, ferritin, transferrin saturation, Ret-Hb, RDW, and serum zinc).

Validated questionnaires will be used to assess:

* General health-related quality of life (SF-12)
* Postpartum depression (EPDS)
* Restless legs syndrome (IRLS)
* Nutrition and supplement intake
* Birth experience (SCIB) The primary aim is to validate the diagnostic performance of non-invasive ZnPP measurements as a screening tool for iron deficiency in pregnancy. Receiver operating characteristic (ROC) analysis will be conducted to compare non-invasive measurements with expert opinion diagnoses and blood-based markers. Secondary outcomes include the relationship between iron deficiency and maternal fatigue, mood disorders, pregnancy outcomes, and neonatal parameters.

Study Design

* Type: Observational (Longitudinal Cohort)
* Duration per participant: Up to 12 months
* Estimated Enrollment: 500 participants
* Timepoints: 1st, 2nd, 3rd trimester, peripartum, and 60-90 days postpartum
* Location: University Hospital Würzburg, Germany

Eligibility Criteria

Inclusion Criteria:

* Pregnant women aged ≥18 years
* Any gestational age or shortly postpartum
* Written informed consent

Exclusion Criteria:

* Previous participation in the study
* Decline of blood sampling for study purposes
* Inability to provide informed consent

Outcome Measures

Primary Outcome:

• Diagnostic performance (ROC/AUC) of non-invasive ZnPP in detecting iron deficiency

Secondary Outcomes:

* Correlation of iron status with quality of life, postpartum depression, and RLS
* Relationship between iron deficiency and pregnancy/neonatal complications

ELIGIBILITY:
Inclusion Criteria:

* any timepoint during or up to 3 months after pregnancy
* age ≥ 18 years
* written informed consent

Exclusion Criteria:

* previous participation in this study
* refusal of blood sampling
* incapacity to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women ≥ 18 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of non-invasive zinc protoporphyrin for the detection of iron deficiency in pregnancy | through study completion, up to 3 months postpartum
  To validate accuracy of non-invasively measured ZnPP for detection of iron deficiency in pregnancy at prespecified timepoints

SECONDARY OUTCOMES:
Influence of iron status on quality of life of pregnant women | through study completion, up to 3 months postpartum
  To evaluate whether iron deficiency has an impact on the risk of impaired quality of life in pregnancy. Questionnaire: Short Form 12 (SF-12)
Influence of iron status on incidence of postpartum depression | through study completion, up to 3 months postpartum
  To evaluate whether iron deficiency has an impact on the risk of postpartum depression. Questionnaire: Edinburgh Postnatal Depression Scala (EPDS)
Influence of iron status on incidence of restless legs syndrome among pregnant women | through study completion, up to 3 months postpartum
  To evaluate whether iron deficiency has an impact on the risk of restless legs syndrome in pregnancy. Questionnaire: International Restless Legs Scale (IRLS)
Influence of iron status on incidence of preterm birth | peripartum ( about 20 weeks of pregnancy until approximately 6 weeks after delivery. )
  To evaluate whether iron deficiency has an impact on the risk of preterm delivery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Würzburg, Würzburg, Bavaria, Germany